CLINICAL TRIAL: NCT05519540
Title: A Single-dose, Open-label, Single Arm Study to Investigate PK of Xevinapant (Debio 1143) and Its Metabolite, D-1143-MET1 in Healthy East Asian Participants
Brief Title: PK Study of Xevinapant (Debio 1143) in Healthy East Asian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MS202359_0004; 2022-002182-15 (EudraCT Number)
Record Dates: First submitted 2022-08-25; First posted 2022-08-29 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2024-07

CONDITIONS: Healthy
Keywords: East Asian; Japanese; Pharmacokinetic; Ethnic sensitivity
MeSH Terms: interventions — N-benzhydryl-5-(2-(methylamino)propanamido)-3-(3-methylbutanoyl)-6-oxodecahydropyrrolo(1,2-a)(1,5)diazocine-8-carboxamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1: Japanese Participants: Xevinapant (Debio 1143) (Experimental): Xevinapant (Debio 1143) was administered in Healthy Japnaese participants at a dose of 200 milligrams (mg), orally under fasted conditions.
  Interventions: Drug: Xevinapant (Debio 1143)
- Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143) (Experimental): Xevinapant (Debio 1143) was administered in Healthy Non- Japanese participants at a dose of 200 mg, orally under fasted conditions.
  Interventions: Drug: Xevinapant (Debio 1143)

INTERVENTIONS:
Drug: Xevinapant (Debio 1143) — All participants (Japanese and non-Japanese) received a single oral dose of 200mg xevinapant (Debio 1143) on Day 1 under fasted condition.

SUMMARY:
The purpose of this study was to evaluate the pharmacokinetics (PK) of Xevinapant (Debio 1143) and its metabolite D-1143-MET1 as well as safety and tolerability of Xevinapant (Debio 1143) in healthy East Asian participants.

ELIGIBILITY:
Inclusion Criteria:

* Healthy participant of Japanese or other East Asian origin. Group 1: Japanese participants must be first generation (born in Japan) with both biological parents and all 4 biological grandparents being Japanese native born, lived for less than (<)10 years outside of Japan, and have no significant change in lifestyle since leaving Japan. Group 2: Other non-Japanese East Asian participants must have both biological parents and 4 biological grandparents of East Asian descent, lived for <10 years outside of their countries, and have no significant change in lifestyle since leaving from there. East Asia includes Korea or Greater China
* Overtly healthy participants as determined by medical evaluation, including medical history, physical examination, laboratory tests, and cardiac monitoring (blood pressure, heart rate, and 12-lead resting ECG)
* Have a body weight within 50 and 110 kilograms [kg] (inclusive) and Body Mass Index (BMI) within the range 18.0 to 32.0 kilograms per meter square [Kg/m^2] (inclusive)
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* History of clinically relevant disease of any organ system that may interfere with the objectives of the study or provide a risk to the health of the participant
* History of relevant drug hypersensitivity, ascertained or presumptive allergy/ hypersensitivity to the active drug substance and/or formulation ingredients history of serious allergic reactions leading to hospitalization or any other allergy reaction in general, which the Investigator considers may affect the safety of the participant and/or outcome of the study
* Ongoing or active clinically significant viral (including Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2)), bacterial or fungal infection, or any major episode of infection requiring hospitalization or treatment with parenteral anti-infectives less than or equal to (<=) 4 weeks prior to or during Screening Period, or completion of oral anti-infectives <= 2 weeks prior to Screening Visit. Vaginal candidiasis, onychomycosis, and genital or oral herpes simplex virus considered to be sufficiently controlled will not be exclusionary
* History of splenectomy
* History of any malignancy (hematologic or solid tumor) before the Screening Visit, except for adequately treated superficial basal cell carcinoma of the skin (no more than 3 lesions requiring treatment in lifetime) or carcinoma in situ/cervical intraepithelial neoplasia of the uterine cervix
* History of or a positive screening test for hepatitis B, hepatitis C, or human immunodeficiency virus type I and II
* Use of any investigational drug in any clinical study within 5 half-lives from last administration
* Other protocol defined exclusion criteria could apply

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2022-09-26 (Actual); Primary Completion 2023-04-21 (Actual); Study Completion 2023-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck Healthcare KGaA, Darmstadt, Germany, an affiliate of Merck KGaA, Darmstadt, Germany
Locations (1):
- Labcorp Clinical Research Unit Limited, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No
We are committed to enhancing public health through responsible sharing of clinical trial data. Following approval of a new product or a new indication for an approved product in both the US and the European Union, the study sponsor and/or its affiliated companies will share study protocols, anonymized patient data and study level data, and redacted clinical study reports with qualified scientific and medical researchers, upon request, as necessary for conducting legitimate research. Further information on how to request data can be found on our website bit.ly/IPD21

REFERENCES:
- See also: Trial Awareness and Transparency website — https://clinicaltrials.emdgroup.com/en/trial-details/?id=MS202359_0004
- See also: Medical Information Location Map - Med Info Contacts — https://www.merckgroup.com/en/company/contact-us/medinfo-contact-map.html

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 47 participants were screened, of which 24 participants (12 Japanese participants and 12 non-Japanese East Asian participants) were enrolled in the study.
Period: Overall Study
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143) | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (7.1) | 29 (6.6) | 30 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 12 | 12 | 24
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 12 | 12 | 24
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Sample Time (AUC0-tlast) of Xevinapant (Debio 1143)
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to the last sampling time (tlast) at which the concentration is at or above the lower limit of quantification. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: The Pharmacokinetics (PK) Analysis Set included all participants who received at least one dose of study intervention and provided at least one measurable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours*nanogram per milliliter (h*ng/mL) | 9780 (34.6) | 10200 (21.4)

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Xevinapant (Debio 1143)
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at t last , as estimated using the linear regression from Terminal first order (elimination) rate constant (Lambda z) determination. AUC0-inf = AUC0-t plus Clast pred/lambda z. Lambda Z was terminal elimination rate constant determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: The PK Analysis Set included all participants who received at least one dose of study intervention and provided at least one measurable postdose concentration.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
h*ng/mL | 9860 (34.4) | 10200 (21.3)

3. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Xevinapant (Debio 1143)
Description: Cmax was obtained directly from concentration versus time curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
ng/mL | 2070 (35.6) | 2160 (32.9)

4. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious TEAEs, and Related TEAE's
Description: An Adverse event (AE) was defined as any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease associated with the use of study drug, whether or not considered related to the study drug or worsening of pre-existing medical condition, whether or not related to study drug. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. An AE was considered as 'treatment emergent' if it occurred after the first drug administration of each period or if it was present prior to drug administration but exacerbated after the drug administration. TEAEs included both serious TEAEs and non-serious TEAEs.
Time Frame: Up to Day 8
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
Participants
  TEAEs | 3 | 5
  Serious TEAE | 0 | 0
  Related TEAE's | 2 | 1

5. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs) by Severity
Description: Severity of TEAEs were graded using Qualitative Toxicity Scale, as follows: Mild: Participant is aware of the event or symptom, but the event or symptom is easily tolerated; Moderate: Participant experiences sufficient discomfort to interfere with or reduce his or her usual level of activity; Severe: Significant impairment of functioning: the participant is unable to carry out his or her usual activities. Number of participants with TEAEs by severity were reported.
Time Frame: Baseline (Day 1) up to Day 8
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
Participants
  Mild TEAEs | 3 | 4
  Moderate TEAE | 0 | 1
  Severe TEAE's | 0 | 0

6. Secondary Outcome: Number of Participants With Clinically Significant Changes From Baseline in Laboratory Values
Description: The laboratory measurements included hematology, blood chemistry and urinalysis. Number of participants with clinically significant changes from baseline in laboratory values were reported. Clinically Significance was decided by investigator.
Time Frame: Baseline (Day 1) up to Day 8
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
Participants
  Hematology | 0 | 0
  Biochemistry | 0 | 0
  Urinalysis | 0 | 0

7. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in 12-lead Electrocardiogram (ECG) Findings
Description: The 12-lead ECG recordings were obtained after 5 minutes of rest in a semi-supine position. ECG recordings included rhythm, ventricular rate, PR interval, QRS duration, QT and QTc intervals. Number of participants with clinically significant changes from baseline in 12-lead ECG findings were reported. Clinically significance was decided by investigator.
Time Frame: Baseline (Day 1) up to Day 8
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

8. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital sign assessment included blood pressure, pulse rate, body temperature and respiration rate. Number of participants with clinically significant changes from baseline in vital signs were reported. Clinically significance was decided by investigator.
Time Frame: Baseline (Day 1) up to Day 8
Population: The safety analysis set included all participants who were administered any dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

9. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of Xevinapant (Debio 1143)
Description: AUC0-24 is defined as the area under the concentration-time curve (AUC) from time zero (= dosing time) to 24 hours. AUC0-24 was calculated using the mixed log-linear trapezoidal rule.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
h*ng/mL | 9160 (34.3) | 9460 (20.6)

10. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Xevinapant (Debio 1143)
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours | 0.750 [0.500 to 2.50] | 1.00 [0.500 to 1.50]

11. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Xevinapant (Debio 1143)
Description: t1/2 was the time measured for the concentration to decrease by one half. Terminal half-life calculated by natural log 2 divided by lambda z. Terminal first order (elimination) rate constant was determined from the terminal slope of the log-transformed concentration curve using linear regression on terminal data points of the curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours | 9.38 (21.2) | 10.5 (28.7)

12. Secondary Outcome: Apparent Clearance (CL/f) of Xevinapant (Debio 1143)
Description: The apparent total body clearance of study intervention following extravascular administration, taking into account the fraction of dose absorbed. CL/f was calculated as Dose/AUC0-inf, where AUC0-inf was estimated by determining the total area under the curve of the concentration versus time curve extrapolated to infinity. AUC0-inf was calculated as AUC0-t + Clast pred/Lambda Z, where Clast pred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the lower limit of quantification (LLQ) and Lambda Z was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter per hour
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
liter per hour | 20.3 (34.4) | 19.6 (21.3)

13. Secondary Outcome: Apparent Volume of Distribution During Terminal Phase (Vz/f) of Xevinapant (Debio 1143)
Description: The apparent volume of distribution during the terminal phase following extravascular administration, based on the fraction of dose absorbed. For single dose Vz/f = Dose/(AUC0-inf*Lambda Z), where AUC0-inf = (AUC0-t + Clast pred/Lambda Z). Clastpred was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLQ and Lambda Z = the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
liter | 274 (36.1) | 296 (27.6)

14. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Measurable Concentration (AUC0-t Last) of Metabolite D-1143-MET1
Description: as for outcome 1
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours*nanogram per milliliter (h*ng/mL)
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours*nanogram per milliliter (h*ng/mL) | 13800 (28.3) | 14400 (34.1)

15. Secondary Outcome: Area Under Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24) of Metabolite D-1143-MET1
Description: The area under the concentration-time curve (AUC) from time zero (= dosing time) to 24 hours. Calculated using the mixed log-linear trapezoidal rule (linear up, log down).
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
h*ng/mL | 13000 (27.4) | 13400 (31.7)

16. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero Extrapolated to Infinity (AUC0-inf) of Metabolite D-1143-MET1
Description: The AUC from time zero (dosing time) extrapolated to infinity, based on the predicted value for the concentration at t last , as estimated using the linear regression from Terminal first order (elimination) rate constant (Lambda z) determination.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: h*ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
h*ng/mL | 13800 (28.2) | 14500 (34.1)

17. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Metabolite D-1143-MET1
Description: Cmax was obtained directly from concentration versus time curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
ng/mL | 1240 (22.2) | 1240 (21.5)

18. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of Metabolite D-1143-MET1
Description: Tmax was obtained directly from the plasma concentration versus time curve.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours | 3.00 [2.00 to 4.00] | 3.00 [2.50 to 4.00]

19. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Metabolite D-1143-MET1
Description: as for outcome 11
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
hours | 5.23 (17.3) | 7.30 (54.4)

20. Secondary Outcome: Metabolite-to-parent Molar Ratio for AUC0-t (MR_AUC0-t) of Xevinapant and D-1143-MET1
Description: AUC0-tlast Molar Ratio is the ratio of AUC0-t molar values of the metabolite compared to the parent calculated by dividing AUC0-t molar values of metabolite D-1143-MET1 with those of xevinapant.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
ratio | 1.66 (40.9) | 1.68 (31.7)

21. Secondary Outcome: Metabolite-to-parent Molar Ratio for AUC0-inf (MR_AUC0-inf) of Xevinapant and D-1143-MET1
Description: AUC0-inf last Molar Ratio is the ratio of AUC0-inf molar values of the metabolite compared to the parent calculated by dividing AUC0-inf molar values of metabolite D-1143-MET1 with those of xevinapant.
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
ratio | 1.65 (40.5) | 1.67 (31.6)

22. Secondary Outcome: Metabolite-to-parent Molar Ratio for Cmax (MR_Cmax) of Xevinapant and D-1143-MET1
Description: Cmax Molar Ratio is the ratio of cmax molar values of the metabolite compared to the parent calculated by dividing Cmax molar values of metabolite D-1143-MET1 with those of xevinapant
Time Frame: Predose, 0.25, 0.5, 1.0, 1.5, 2, 2.5, 3, 4, 6, 8, 12, 24 , 36, 48 and 72 hours postdose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
Number analyzed (Participants) | 12 | 12
ratio | 0.704 (42.7) | 0.679 (31.7)

ADVERSE EVENTS:
Time Frame: Up to Day 8
Arm/Group | Group 1: Japanese Participants: Xevinapant (Debio 1143) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 5/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1: Japanese Participants: Xevinapant (Debio 1143) (N=12) | Group 2: Non-Japanese East Asian Participants: Xevinapant (Debio 1143) (N=12)
Retching (Gastrointestinal disorders) | 0 (0) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 1 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-06-10): https://cdn.clinicaltrials.gov/large-docs/40/NCT05519540/Prot_000.pdf
  • Statistical Analysis Plan (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/40/NCT05519540/SAP_001.pdf